CLINICAL TRIAL: NCT06985628
Title: Alleviating Dyspnea With Non-Invasive Neuromodulation : A Feasibility Sham-Controlled Randomized Trial
Brief Title: Alleviating Dyspnea With Non-Invasive Neuromodulation
Acronym: PNEURO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Association Pulmonaire du Quebec (Other); Fonds de la Recherche en Santé du Québec (Other Government); Québec Air-Intersectorialité-Respiratoire-Son network (Unknown)
Responsible Party: Principal Investigator, Simon Couillard, M.D. M.Sc., Assistant-professor in medicine, Respirology Service, Department of Medicine, Université de Sherbrooke
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-5604
Record Dates: First submitted 2024-08-15; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Dyspnea; Chronic Obstructive Pulmonary Disease Severe
Keywords: Dyspnea; Breathlessness; Neuromodulation; Transcutaneous electrical nerve stimulation (TENS); Vagal nerve stimulation (VNS); Trigeminal nerve; Chronic obstructive pulmonary disease (COPD); Cardiopulmonary exercise test (CPET)
MeSH Terms: conditions — Dyspnea; Pulmonary Disease, Chronic Obstructive | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: At visit 1, participants will be randomized to one of four schedules for subsequent study procedures: VNSsa (visit 1 sham → visit 2 active), VNSac (visit 1 active → visit 2 sham), TENSsa (visit 1 sham → visit 2 active), or TENSac (visit 1 active → visit 2 sham) in a 1:1:1:1 ratio through the randomization function of REDCap.
  VNS : Vagal nerve stimulation TENS : Transcutaneous electrical nerve stimulation
Who Masked: Participant
Masking Description: This study employs a single-blinded format, where participants are unaware if they are receiving the sham or the real interventions, but the researchers in charge of data collection or of the analysis are not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- tVNS (Experimental): Two options of schedule (according to crossover randomization):
  - VNSsa : Visit 1 : sham → Visit 2 : active tVNS
  - VNSac : Visit 1 : active tVNS → Visit 2 : sham
  Interventions: Device: Transcutaneous vagal nerve stimulation (tVNS)
- Trigeminal TENS (Experimental): Two options of schedule (according to crossover randomization):
  - TENSsa : Visit 1 : sham → Visit 2 : active trigeminal TENS
  - TENSac : Visit 1 : active trigeminal TENS → Visit 2 : sham
  Interventions: Device: Transcutaneous electrical nerve stimulation (TENS)

INTERVENTIONS:
Device: Transcutaneous vagal nerve stimulation (tVNS) — tVNS will be applied at the cervical level of the vagal nerve.
  Other Names: gammaCore
  Arms: tVNS
Device: Transcutaneous electrical nerve stimulation (TENS) — TENS will be applied facially on the trigeminal nerve.
  Arms: Trigeminal TENS

SUMMARY:
The goal of this feasibility sham-controlled randomized trial is to assess the feasibility of studying non-invasive neuromodulation techniques, specifically transcutaneous vagal nerve stimulation (tVNS) and transcutaneous electrical nerve stimulation (TENS) of the trigeminal nerve to alleviate dyspnea in patients with chronic pulmonary disease.

The main question it aims to answer is:

Despite challenges in dyspnea generation and measurement, could non-invasive neuromodulation be reliably studied in chronic obstructive pulmonary disease (COPD) with severe dyspnea?

Researchers will compare tVNS and trigeminal TENS to a sham (where the device is applied, but without stimulation) in order to see if non-invasive neuromodulation could relieve dyspnea.

At the time of rehabilitation pre-assessment, participants routinely undergo a baseline maximal Cardiopulmonary Exercise Testing (CPET) on ergocycle to measure VO2max with repetitive assessments of the Borg scale and continuous monitoring of vital signs (oxygen saturation, heart rate, blood pressure, respiratory rate) throughout the test. Spirometry and symptom questionnaires (CAT score) are also routinely measured. In two dedicated study visits conducted 2 weeks apart from each other, n=8 participants will perform a submaximal constant workrate (CRW) at 80% workload of the VO2 max, either with cervical tVNS (n=4) or trigeminal TENS (n=4). In a cross-over design, both patient groups will undergo sham and active treatment of the neuromodulation technique in a randomly assigned number.

DETAILED DESCRIPTION:
Objectives

Primary objective:

- To assess the feasibility of studying non-invasive neuromodulation techniques, specifically cervical transcutaneous vagal nerve stimulation (tVNS) and trigeminal transcutaneous electrical nerve stimulation (TENS) of the trigeminal nerve to alleviate dyspnea in patients with severe chronic pulmonary disease.

Exploratory objectives:

* To evaluate alterations in dyspnea perception resulting from the interventions.
* To review the involvement of trigeminal and vagal nerves in the neurological pathways of dyspnea, as documented in existing scientific literature.
* To evaluate the convenience of VNS and TENS devices and of their use on the patients with chronic pulmonary diseases.
* To assess the quality of the sham employed in this trial.

METHODS

Study design

We propose an observational, prospective, feasibility, cross-over trial to explore the potential of two non-invasive neuromodulation methods, tVNS and trigeminal TENS, to alleviating dyspnea. The study protocol follows the SPIRIT (Standard Protocol Items: Recommendations for Interventional Trials) guidelines. This study employs a single-blinded format, where participants are unaware if they are receiving the sham or the real interventions, but the researchers in charge of data collection or of the analysis are not blinded. The study will be conducted at the Centre Hospitalier Universitaire de Sherbrooke (CHUS)'s research centre, and participants will be selected from the chronic obstructive pulmonary disease (COPD) pulmonary rehabilitation clinic at CHUS, in Quebec, Canada.

Research metrics

Although this is a feasibility study focusing on recruitment, retention, adverse effects, and acceptability (using a Likert questionnaire), our overarching research aims to explore the impact of dyspnea in individuals by using the submaximal Constant work rate (CWR) at 80% of VO2max to experimentally provoke dyspnea symptoms and evaluate the effects of our proposed relieving techniques. Spirometry according to American Thoracicy Society 2019 standards will be employed to evaluate pulmonary function, encompassing key parameters such as Forced Expiratory Volume in 1 second (FEV1), Forced Vital Capacity (FVC), and FEV1/FVC. This spirometry will be done without holding inhalers (i.e. "on-treatment spirometry" : patient will be instructed to take their inhalers that morning). Basic vital signs, including oxygen saturation, heart rate, arterial blood pressure, respiratory rate and temperature, will also be measured to ensure the safety of the patients and to support the study. Subjective dyspnea assessments will be carried out using the Borg scale (0-10), a 100mm Visual analogue scale (VAS) for dyspnea, complemented by the Modified Medical Research Council (mMRC) dyspnea scale for individuals with COPD, the COPD Assessment Test (CAT), and the time to return to initial Borg Score serves as a measure of recovery following the exercise test. Data on rehabilitation performance will include measurements of workload, VO₂ max, pedaling time, and breathing and cardiac reserves. To confirm (yes or no) whether the baseline visit reached maximal effort at VO2max, the criteria for maximal effort from the ERS statement on the standardisation of cardiopulmonary exercise testing in chronic lung diseases will be applied. The quality of blinding with the proposed sham will also be assessed. Common short-term side effects will be assessed frequently, with a minimum of one evaluation at the end of each experimental visit using a standardized questionnaire designed for the interventions of the study. This approach aims to promptly identify and screen for any undesirable effects experienced by participants. Other questions will assess participants' expectations and perceived intervention efficacy during each exercise test using a numeric analogue scale (NAS). A short questionnaire will evaluate the anxiety, depression, and catastrophization related to breathlessness. The St George's Respiratory Questionnaire (SGRQ) will be used to assess participants' initial quality of life status.

Schedule of visits

Throughout the entire duration of the study, participants' complete medication regimen will be assessed, and their medication must remain stable during the trial. As part of the pulmonary rehabilitation program, the eight participants will undergo a medically advised first cardiopulmonary exercise testing (CPET) at VO2max following the data measurement procedures of a standard medical visit. The Borg scale will be evaluated before the test, every 3 minutes during the test, at end of test. For the baseline visit, only SpO2 will be measured before and after CWR. Additionally, spirometry parameters, including FEV1, FVC, and FEV1/FVC will be measured before the test. Data on rehabilitation performance, such as VO2 max, breathing and cardiac reserve, and the assessment of maximal effort testing, will be useful for the setting of the next two visits. This baseline CWR is crucial as it accounts for the effects of adaptation to the physical test (learning effect), ensuring that any observed changes in subsequent tests are not merely due to physiological adaptations or normal variations that occur in every test conducted under this protocol.

At least two weeks later, participants undergo a submaximal CWR at 80% of VO2max and with the same data measurement of the baseline CWR with the addition of more dyspnea evaluation questionnaires. At the beginning of the visit, demographic data and medical records (confirmed via data entry form), the SGRQ, and the Psychological Components Questionnaire (PCQ) will be administered. These include the Borg scale assessed every minute during the test, the mMRC and CAT questionnaires administered before the test, and the VAS recorded before and after CWR. Participant's expectations regarding the efficacy of the intervention will be assessed at rest, both with and without stimulation. At the end of the protocol, stimulation and perceived efficacy will be evaluated to gather additional subjective data on relief perception and the quality of the sham. Additionally, the time taken to return to the initial Borg score at rest following CWR will be measured. Vital signs, including oxygen saturation (O2), heart rate (HR), blood pressure (BP), respiratory rate (RR), temperature (T˚) will also be monitored throughout the entire duration of the test (T˚ that are only assessed before CWR). Participants will at this point receive either a cervical or facial neurostimulator, delivering cervical transcutaneous vagal nerve stimulation (tVNS) or trigeminal transcutaneous nerve stimulation (TENS). The tVNS GammaCore device operates with predefined parameters, delivering a 5000-Hz pulse at a frequency of 25 Hz, while stimulation intensity remains adjustable. For TENS, the initial settings could involve a 60-microsecond pulse duration at a frequency of 100 Hz. The intensity can be modulated and these parameters may be adjusted during preliminary tests of the devices and for each patient as needed. However, the effectiveness threshold, related to pain modulation, in terms of amplitude of the electrostimulation, depends on the patient. Then, for both tVNS and trigeminal TENS, the amplitude will be adjusted to reach a threshold where the patient perceives a strong stimulation, experiencing paresthesia on the trigeminal area, while remaining comfortable for them. For the sham TENS and tVNS, we suggest informing patients that two different modes of stimulation will be used, one of which will feel stronger than the other. This allows us to activate the device during the intervention and adjust it to a level where the skin experiences a mild tingling sensation or even to turn off the device for the sham condition. This stimulation will remain below the threshold of the gate control theory, being clinically ineffective. Then, the sham is conceptualized using the same device (TENS or tVNS) for both experimental visits. For both the sham and intervention, light and sound confounding stimuli on the devices will be used to enhance blinding efficiency and minimize the placebo effect in our comparative analysis.

Resulting from a informatic random attribution, 4 participants receive cervical tVNS (gammaCore Sapphire D Device, electroCORE inc.: approved by Health Canada, see 'Feasibility') and 4 participants receive trigeminal TENS, applied by a specialized physiotherapist. In each group, 2 participants initially receive the intervention while 2 participants receive the sham.

Two weeks after the first experimental visit, those who received an intervention (tVNS or trigeminal TENS) will receive the sham, and those who received the sham will receive an intervention. This switch occurs according to the randomization process of the crossover group assignment. They all undergo a final submaximal CWR with the same data collected sequence as for the first experimental visit two weeks ago.

In case of technical issues or other concerns affecting the validity of the test or the data collected during one of the visits, an additional visit (at week 4) could be added after the last experimental visit. If this visit takes place, it will follow the same exercise testing and intervention protocols as the two preceding experimental visits.

If patients experience significant discomfort or adverse effects during the test or interventions, they should immediately inform the healthcare provider so that appropriate measures can be taken to reassure and manage the patient effectively, including possibly stopping the procedure if necessary. Otherwise, the standardized questionnaire specific for this study will be applied by the investigators at the end of every visit. During visits, respiratory therapist will be present to evaluate and supervise pulmonary rehabilitation exercise tests. A pulmonologist will be available in case of any major medical issues. Study visits will be completed before starting rehabilitation. Rehabilitation program typically begins within 5 months of the initial medically recommended visit (Baseline Visit).

Data and sample management

Demographic and medical-record data regarding patients will be collected for patient enrollment based on inclusion and exclusion criteria, and to analyze correlations between feasibility outcomes and patient characteristics. This data will only be accessible through specific computers with authorized permission to access the ARIANE system at CHUS. Throughout each data collection session for the study's tests, comprehensive notes will be written manually on paper clinical notes, and standardized scales and clinical research forms will be completed by hand. The data will then be transcribed into a REDCap® project for optimized data management. No data monitoring committee (DMC) was deemed necessary, as the risks associated with the study's non-invasive procedures are considered minimal. The interventions, tVNS and TENS, involve clinically approved devices with a well-established safety profile and no significant risk.

Statistical analyses

Descriptive analysis will be conducted for the primary objectives to evaluate the feasibility parameters. For the exploratory objective concerning the alteration in dyspnea perception and pulmonary parameters, several statistical methods will be employed. The Borg slope will be analyzed using a linear mixed model, which accounts for both fixed and random effects, allowing for the evaluation of changes over time within individuals. Paired sample T-tests will compare parameters before and after the interventions, determining if there is a significant difference. The chi-square test will assess the association between categorical variables.

ELIGIBILITY:
Inclusion Criteria:

* Severe COPD (between FEV1 20-50%, FEV1/FVC < 0.7, and smoking history of ≥ 10 pack-years, 3rd-4th grade on the dyspnea scale modified Medical Research Council (mMRC), COPD Assessment Test (CAT) score ≥ 10)
* Significant chronic dyspnea for at least 6 months
* Referred for pulmonary rehabilitation
* Physical capability to undergo submaximal constant work rate (CRW)
* Ability to comprehend the implications of the procedures and follow-up visits and provide free informed consent

Exclusion Criteria:

* Presence of concurrent pulmonary restrictive features
* Neurological disorders susceptible to be influenced by neurostimulation procedures, including epilepsy, Parkinson's disease, trigeminal neuralgia, dysautonomia, and vagal disorders
* Unstable arrhythmias, and other cardiac instabilities
* Patients with cardiac pacemakers, defibrillators, or other metal implants
* Patients who have undergone pulmonary resection resulting in the absence of pulmonary lobe(s) or complete lung
* Other serious dyspneic conditions, such as anemia, heart failure with decreased ejection fraction, or mitochondrial dysfunction
* Pregnancy
* Active infections
* Known reactions or intolerance to tVNS or trigeminal TENS

Patients must have no moderate-to-severe exacerbations (defined as an increase in symptoms for more than 3 days requiring corticosteroids or antibiotics, or hospitalisation) for at least one month before the baseline visit and at least one month before the first experimental visit (W0 visit). Participants that were randomized yet experience an exacerbation between the first (at week 0) and second (at week 2) experimental visits will be removed from the trial.

*Abbreviations : COPD : chronic obstructive pulmonary disease FEV1 : Forced Expiratory Volume in one second FVC : Forced vital capacity tVNS : Transcutaneous vagal nerve stimulation TENS : Transcutaneous electrical nerve stimulation

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Sample study completion proportion | At every visit until the visit 2 (at week 2)
  Percentage of recruited patients attending all visits and completing all tests

SECONDARY OUTCOMES:
General acceptability of the study procedures (exercise testing and interventions) | At the end of the visit 2 (at week 2)
  It will be assessed by a Likert score (0-45 points equally divided on 9 questions regarding : effectiveness, impact, safety, side effects, acceptability, compliance, accessibility, awareness, and importance of the interventions).
Recruitment results | At the visit 1 (at week 0)
  Percentage of recruited patients on the target sample size, which is 2 x n=4
Adverse effects and undesirable events regarding the study procedures (exercise testing and interventions) | At every visit until the visit 2 (at week 2)
  Qualitative listing using systematically an adaptation of the Common Terminology Criteria for Adverse Events (CTCAE) 5.0.1.
Occurrence of any adverse effects and undesirable events | At every visit until the visit 2 (at week 2)
  Quantitative statistical assessment of specific adverse events (relative risk, timing of occurence during the experimentation, etc.)
Change from baseline for each intervention (tVNS and trigeminal TENS) | At every visit until the visit 2 (at week 2)
  Absolute change from baseline to maximum modified Borg Rating Of Perceived Exertion score (score : 0 to 10 ; Minimal clinically important difference (MCID)=1) and Borg score slope during test (measured every minute during constant work rate (CWR)) for each intervention (tVNS, transcutaneous vagal nerve stimulation, and TENS, transcutaneous electrical nerve stimulation).
Absolute change in pedaling time at the same pace from baseline | At every visit until the visit 2 (at week 2)
Sham evaluation | At the end of the visit 2 (at week 2)
  Blinding assessment of the sham will be based on expectation and efficacy-related questions during study visits, along with a dedicated sham questionnaire designed to evaluate participants' ability to distinguish the sham from the active intervention, in order to assess the potential impact of unblinding on the scientific evaluation of intervention efficacy, particularly in relation to placebo effect considerations in neuromodulation trials.

CONTACTS AND LOCATIONS:
Overall Officials: Joël St-Pierre, MD MSc candidate, Principal Investigator — Université de Sherbrooke; Simon Couillard, MD MSc, Study Director — Université de Sherbrooke; Christian Iorio-Morin, MD PhD, Study Director — Université de Sherbrooke
Locations (1):
- Centre hospitalier universitaire de Sherbrooke (CHUS), Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data of this study may be shared if the investigators proposed use of the data has been approved by the study principal investigator and an institutional research ethics committee.
Time Frame: Up to 2035
Access Criteria: Data of this study may be shared if the investigators proposed use of the data has been approved by the study principal investigator and an institutional research ethics committee.

REFERENCES:
- [Derived] St-Pierre J, Mailhot-Larouche S, Garand G, Vezina FA, Leonard G, Iorio-Morin C, Couillard S. Non-invasive neuromodulation for alleviating dyspnoea: protocol for a feasibility sham-controlled randomised trial. BMJ Open. 2025 Jul 22;15(7):e103891. doi: 10.1136/bmjopen-2025-103891. PMID 40701604